CLINICAL TRIAL: NCT01111097
Title: Phase 1, Open-Label, Single-Arm, Clinical and Metabolomics Study of Dichloroacetate (DCA) in Adults With Recurrent Malignant Brain Tumors
Brief Title: Study of the Safety and Efficacy of Dichloroacetate (DCA) in Glioblastoma and Other Recurrent Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-2010; CTSI (Other: Ocala Dames); UL1TR000064 (NIH)
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Brain Tumor; Glioblastoma
Keywords: Brain tumors, Glioblastoma and DCA; Brain tumor,Glioblastoma recurrent
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Subjects are given a dose of Dichloroacetate 4mg/kg twice a day for 30 days
  Interventions: Drug: Dichloroacetate
- Cohort 2 (Active Comparator): Subjects are given a dose of Dichloroacetate 12.5mg/kg twice a day for 30 days
  Interventions: Drug: Dichloroacetate

INTERVENTIONS:
Drug: Dichloroacetate — Subjects after passing the inclusion criteria are given a dose of dichloroacetate 4mg/kg bid for thirty days. While in the clinical research center they participate in a breath test where they exhale through a straw into a glass tube. This will measure CO2. They are monitored every two weeks for side effects and return to the clinical research center for evaluation in thirty days. They undergo another breath test and if all health parameters are within normal limits they are given a month's supply of dichloroacetate. The cycles continue unless a serious adverse event occurs or the PI judges the side effects preclude another 30 days of medication
  Other Names: DCA

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of oral Dichloroacetate (DCA) in the treatment of recurrent malignant brain tumors (RMBTs). RMBTs are defined as either: 1) malignant tumors, originating in the brain, that have recurred at least once or 2) malignant tumors originating elsewhere in the body that have spread to the brain at least once. Otherwise, there are no limitations to the number of prior recurrences. There are no limitations to the number or types of prior therapies.

DETAILED DESCRIPTION:
Malignant brain tumors are defined as any World Health Organization grade III-IV glioma and any solid tumor metastasis (spread) to the brain. Recurrent malignant brain tumors (RMBTs) are defined as either: 1) malignant tumors, originating in the brain, that have recurred at least once or 2) malignant tumors originating elsewhere in the body that have spread to the brain at least once. They share an increasing incidence, clinical and radiographic characteristics, lack of effective therapies, tendency to recur, and poor outcome. Importantly, recurrent malignant brain tumor's shared characteristics may be usefully exploited by an emerging class of biologic agents called metabolic modulators of which Dichloroacetate (DCA) is the drug in the class most thoroughly investigated clinically. DCA's mechanism of action and tolerability have been extensively demonstrated in the treatment of chronic metabolic disorders. Furthermore, the preciseness of DCA's mechanism of action appears to target abnormal tumor cell metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to consent for self. Subject must have either:

  1. a brain metastasis or
  2. a WHO III-IV glioma that has recurred at least once. Females of child bearing age must have (-) pregnancy test.
* Females of child bearing age must use birth control while in study.
* Adequate organ function as determined by laboratory testing.
* Absence of peripheral neuropathy of moderate or greater severity (physician determined).
* Greater than 4 weeks time from previous anti-neoplastic (anti-cancer) therapy.
* Subject must have a Karnofsky Performance Status (KPS) of greater than or equal to 60.
* Subject must have an ECOG performance status of less than or equal to 2.
* There are no limitations to the number of prior recurrences.
* There are no limitations to the number or types of prior therapies.

Exclusion Criteria:

* Medical contraindication for magnetic resonance imaging (MRI)testing.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of DCA in RMBTs. | Within 28 days of starting DCA +/- 3 days
  Oral DCA will be administered until intolerance, toxicity, radiographic progression, or death. Safety and tolerance will be assessed by reviewing available standardized clinical, radiographic, and quality of life (QOL) criteria. The safety and tolerance will also be assessed by reviewing available plasma, urine, and brain tumor tissue for metabolites of the tumor and the effects of DCA thereon.

SECONDARY OUTCOMES:
Conduct an exploratory investigation of the metabolites of patients with RMBTs and the effects of DCA thereon. | One year
  We postulate that the metabolism of RMBTs and the effects of DCA thereon will help investigators understand RMBTs, how DCA works on them, and how to design future treatment studies.

CONTACTS AND LOCATIONS:
Overall Officials: Erin M. Dunbar, MD, Principal Investigator — University of Florida; Peter W. Stacpoole, PhD, MD, Study Chair — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Dunbar EM, Coats BS, Shroads AL, Langaee T, Lew A, Forder JR, Shuster JJ, Wagner DA, Stacpoole PW. Phase 1 trial of dichloroacetate (DCA) in adults with recurrent malignant brain tumors. Invest New Drugs. 2014 Jun;32(3):452-64. doi: 10.1007/s10637-013-0047-4. Epub 2013 Dec 3. PMID 24297161